CLINICAL TRIAL: NCT05232448
Title: The Effect of Cognitive Behavioral Therapy Education to Elderly Care Students on Ageism, Attitudes to Elderly, Empathy and Body Image
Brief Title: The Effect of Cognitive Behavioral Therapy Education to Elderly Care Students on Outcome Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 210038
Record Dates: First submitted 2022-01-08; First posted 2022-02-09 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Behavioral Therapy; Ageism
Keywords: Elderly care; Ageism; Cognitive Behavioral Therapy; Empathy
MeSH Terms: conditions — Ageism | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Assesors are blinded to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Data collection forms will be applied to the students in the control group first. They will then continue their normal education.
- Intervention Group (Experimental): Data collection forms will be applied to the students in the intervention group first. Afterwards, cognitive-behavioral therapy training will be implemented as four modules, lasting 1 month in total.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy focuses on challenging and changing cognitive distortions and behaviors, improving emotional regulation and the development of personal coping strategies that target solving current problems.
  Arms: Intervention Group

SUMMARY:
The aim of this study, to examine the effects of cognitive behavioral therapy education to elderly care students on ageism, attitudes towards the elderly, empathy and body image.

DETAILED DESCRIPTION:
Students in the control group will continue their normal education. The students in the intervention group will be given training on ageism, elderly attitude, empathy and body image in the cognitive therapy training, which will be given by a psychological counselor who is an expert in the field and will last for a total of 1 month in four modules.

ELIGIBILITY:
Inclusion Criteria:

* Students who do not have hearing, speech and psychiatric problems that prevent communication
* Students who volunteered to participate in the study

Exclusion Criteria:

- Students who do not want to be involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Kogan Attitudes Toward Old People Scale | Change from Baseline Kogan Score at 1 month
  The scale measures the attitudes of individuals towards the elderly. An increase in the total score indicates that the individual has a positive attitude towards the elderly. 34 is the lowest score, and 204 is the highest score obtained from the scale. A high score obtained from the scale indicates a positive attitude towards older people.
The Cognitive Affective and Somatic Empathy Scales (CASES) for Children | Change from Baseline CASES Score at 1 month
  The scale was developed to evaluate the empathy levels of children and adolescents.The total score for thirty items ranges from 0 to 60, and it is thought that the higher the score, the higher the tendency to empathize.
Ageism Attitude Scale | Change from Baseline Ageism Attitude Scale at 1 month
  It is a scale with three sub-dimensions: limiting the life of the elderly, positive discrimination and negative discrimination attitudes towards the elderly. A high score indicates a positive attitude. The highest possible score from the survey was 190 and the lowest was 38 according to this scoring scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Dovan, BSc, Principal Investigator — Koycegiz District Directorate of Social Services; İsmet Tümtürk, BSc, Principal Investigator — Ege University
Locations (1):
- Muğla Sıtkı Koçman University Vocational School of Health Services, Muğla, Köyceğiz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No